CLINICAL TRIAL: NCT03336658
Title: Assessment of Intratumoral Budding (ITB) in Preoperative Biopsies of Colon and Rectal Cancer Patients: a Prospective Observational Study
Brief Title: Intratumoral Budding (ITB) in Preoperative Biopsies of Colon and Rectal Cancer
Acronym: ITB
Status: Active, not recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 393/14
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: CRC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tumor buds will be Immunohistochemically stained with a pancytokeratin marker
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
All the preoperative biopsies of patients suffering colorectal cancer (CRC) will be immunohistochemically stained with a pancytokeratin marker to detect Tumor buds. then, the intratumoral buds (ITB) in the densest Region of Tumor buds, namely the "hot spot" will be counted. Subsequently, the probability of N stage (lymphnodes), M stage (metastases) and disease free survival (DFS) will be calculated based on an existing logistic Regression model already developed by our previous retrospective work. Additionally, a Standardisation of ITB using a well- established Software will develop an algorithm which will help to eliminate inter- observer variability of Tumor budding Counts.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed stages I and IV colorectal cancer (CRC)
* Age ≥ 18 years
* Written Informed Consent

Exclusion Criteria:

* No consent
* < 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Stages I to IV colorectal cancer
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
correlation of ITB based calculated N stage with real N stage in CRC - patients | 24 months

SECONDARY OUTCOMES:
correlation of ITB based calculated DFS with real DFS in CRC - patients | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Beat Schnüriger, PD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Department of visceral surgery and transplant surgery, Berne University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No